CLINICAL TRIAL: NCT01295385
Title: Contribution Of Nuclear Magnetic Resonance Imaging In The Study Of Diabetic Cardiomyopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-A00233-36; 2009-41
Record Dates: First submitted 2011-01-26; First posted 2011-02-14 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Diabetic; Cardiomyopathy
Keywords: type 2 diabetes; Cardiovascular diseases; coronary syndrome have abnormalities of glucidic metabolism
MeSH Terms: conditions — Cardiomyopathies; Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- healthy volunteers (Experimental)
  Interventions: Other: NUCLEAR MAGNETIC RESONANCE IMAGING
- patients with a diabetic cardiomyopathy (Active Comparator)
  Interventions: Other: NUCLEAR MAGNETIC RESONANCE IMAGING

INTERVENTIONS:
Other: NUCLEAR MAGNETIC RESONANCE IMAGING — Techniques of nuclear magnetic resonance offer interesting perspectives in this context, and particularly to quantify the myocardial blood flow at rest and after "cold pressor test" in a population of healthy volunteers.
  Arms: healthy volunteers
Other: NUCLEAR MAGNETIC RESONANCE IMAGING — Techniques of nuclear magnetic resonance offer interesting perspectives in this context, and particularly to quantify the myocardial blood flow will be obtained by estimating myocardial blood flow at the venous coronary sinus site. This allows us to quantify a possible endothelial dysfunction in a reproducible way. No MRI study in diabetic patients has ever been led until now with this technique and to estimate the metabolic and structural abnormalities in this population.
  Arms: patients with a diabetic cardiomyopathy

SUMMARY:
Diagnosis of diabetic cardiomyopathy is then retained, supposing a change in the coronary microcirculation linked to an endothelial dysfunction. Abnormalities of the myocardial metabolism is frequently associated. It is regrettably about a hypothesis difficult to verify with current medical techniques.This deficiency being not only harmful to the diagnosis, but also to the assessment of the efficiency of the medical treatment on the myocardial metabolism and the endothelial function. Techniques of nuclear magnetic resonance offer interesting perspectives.

DETAILED DESCRIPTION:
These techniques allow in this context:

1. to quantify the myocardial blood flow at rest and after "cold pressor test" in a population of healthy volunteers. The myocardial blood flow will be obtained by estimating myocardial blood flow at the venous coronary sinus site. This allows us to quantify a possible endothelial dysfunction in a reproducible way. No MRI study in diabetic patients has ever been led until now with this technique.
2. to estimate the metabolic and structural abnormalities in this population, with particularly:

   * Quantification of the myocardial metabolism in vivo by spectrometry of phosphorus 31.
   * Structural abnormalities: become integrated into the description of diabetic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old
* patient type 2 diabetes affects taken care more than 5 years to Timone Hospital
* patient with a diabetic cardiomyopathy
* informed and consented

Exclusion Criteria:

* less than 18 years
* Pregnant woman
* patient type 1 diabetes affects
* patient presents a cardiomyopathy mixed (no diabetic)
* patients presents an arrhythmia ventriculaire or above - ventriculaire
* Unstable hémodynamique patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2011-02; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
To quantify the myocardial blood flow at rest and after "cold pressor test" in a population of healthy volunteers | 12 months
  The myocardial blood flow will be obtained by estimating myocardial blood flow at the venous coronary sinus site. This allows us to quantify a possible endothelial dysfunction in a reproducible way. No MRI study in diabetic patients has ever been led until now with this technique.

SECONDARY OUTCOMES:
To estimate the metabolic and structural abnormalities in this population | 12 months
  * Quantification of the myocardial metabolism in vivo by spectrometry of phosphorus 31 which allows to estimate the energy state of the heart by analyzing the phosphorous metabolites with high energy involved in the myocardial energetic metabolism.
  * Structural abnormalities: evaluation of the fibrosis and the collagenic deposits by T1 mapping and measurement of relaxation T2 as well as the study of the late enhancement of gadolinium. These structural abnormalities become integrated into the description of diabetic cardiomyopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Quilici, Doctor, Principal Investigator — APHM
Locations (1):
- Assistance Publique - Hopitaux de Marseille, Marseille, France